CLINICAL TRIAL: NCT06380166
Title: Hepatitis C Lab Testing Comparison Study
Status: Terminated | Type: Observational
Why Stopped: We had difficulty recruiting this population and enrolled only one patient.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Principal Investigator, Ian Gunsolus, Director, Scientific Medical Laboratory, HealthPartners Institute
Other Study IDs: A23-356
Record Dates: First submitted 2024-04-17; First posted 2024-04-23 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to undergo a blood draw
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- In vitro stability investigation
  Interventions: Diagnostic Test: Hepatitis C core antigen

INTERVENTIONS:
Diagnostic Test: Hepatitis C core antigen — Semi-quantitative, automated immunoassay detecting core antigen of hepatitis C virus.

SUMMARY:
Hepatitis C (HCV) HCV antibody assays are the standard of care test used to screen for HCV, but confirmation of acute infection is relegated in the current US guidelines to polymerase chain reaction (PCR) which often takes multiple days and may result in a loss to follow up and treatment, especially in high prevalence populations. HCV core antigen is a new, research use only immunoassay intended for use on the Abbott Alinity i system, an FDA-cleared instrument for clinical chemistry and immunoassay testing. The aim of the study is to evaluate the 48-hour stability of HCV core antigen in fresh serum and plasma specimens collected from individuals with a detectable HCV viral load (HCL VL), as per a recent antibody assay test, under multiple specimen storage conditions mirroring those employed in clinical laboratories.

DETAILED DESCRIPTION:
This study seeks to test the stability of a novel method of hepatitis-C testing called HCV core antigen testing. This will be accomplished by prospectively consenting patients who have had a recent, positive standard of care HCV viral load test, and drawing additional blood to conduct HCV core antigen testing within the infectious period. Viral load amount of the core antigen test will be recorded at baseline and subsequent timepoints. Stability is defined as <10% change from baseline and will be recorded at various timepoints up to 144 hours post-draw. Stability will also be tested at room temperature vs. refrigerated storage and on the gel vs. off the gel processing techniques. This information is necessary to ensure HCV core antigen is sufficiently stable following specimen collection to enable robust, accurate, and precise measurement using the HCV core antigen assay.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Had detectable HCV VL in a standard of care Hepatitis C RNA Quantitative test
* Initial hepatitis C VL testing took place at any HealthPartners lab
* Able to undergo a study blood draw within 3 weeks of initial hepatitis C VL testing
* Ability to sign e-consent prior to presenting for a study lab draw

Exclusion Criteria:

* Age <18 years
* On the HealthPartners research opt-out list
* HCV VL not detectable at follow-up lab draw (screen fail)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have tested positive for Hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Serum on the clot stability | 6 days
  Determine the 48-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at ambient temperatures (20.0-25.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
  Determine the 144-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at refrigerated temperatures (2.0-8.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
Serum off the clot stability | 6 days
  Determine the 48-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at ambient temperatures (20.0-25.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
  Determine the 144-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at refrigerated temperatures (2.0-8.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
Plasma on the gel stability | 6 days
  Determine the 48-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at ambient temperatures (20.0-25.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
  Determine the 144-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at refrigerated temperatures (2.0-8.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
Plasma off the gel stability | 6 days
  Determine the 48-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at ambient temperatures (20.0-25.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.
  Determine the 144-hour reproducibility of HCV core antigen measurements in serum and plasma specimens stored at refrigerated temperatures (2.0-8.0 C) and collected from patients with detectable HCV VLs who completed standard of care Hepatitis C RNA Quantitative testing within the prior 2 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners, Bloomington, Minnesota, United States